CLINICAL TRIAL: NCT03293381
Title: Electrogram-Guided Myocardial Advanced Phenotyping (The eMAP Trial)
Brief Title: Electrogram-Guided Myocardial Advanced Phenotyping
Acronym: eMAP
Status: Terminated | Type: Observational
Why Stopped: As per the investigators decision
Sponsor: University of Pennsylvania (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 826102
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Non-ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: additional biopsies — additional biopsies

SUMMARY:
Fluoroscopy guided EMB and EAM guided EMB on all patients meeting existing guidelines for biopsy.

DETAILED DESCRIPTION:
Non-Ischemic Cardiomyopathy (NICM) is a common cause of heart failure (HF) and death. NICM is a heterogeneous entity, and specific etiologies are infrequently identified. In part due to limited disease characterization, specific treatments are lacking for most of the different underlying causes of NICM. Depending on the cohort, 30-70 percent of patients with new-onset NICM develop persistent systolic dysfunction despite guideline-directed medical therapy, and these patients have high rates of subsequent morbidity and resource utilization.

Current guidelines support the use of endomyocardial biopsy (EMB) in patients with both new-onset and persistent cardiomyopathy. However, EMB is underutilized in these populations due to its low diagnostic yield. A combination of sampling error resulting from standard fluoroscopy-guided EMB in disease entities with patchy myocardial involvement and rudimentary tissue phenotyping of the specimens which are obtained contribute to this low diagnostic yield. In recent years, there has been increasing interest in the use of electro-anatomic mapping (EAM) to help identify areas of myocardium with discrete pathology based on abnormalities in intra-cardiac electrogram voltage and morphologies. Therefore, the primary objective of this protocol is to provide definitive evidence that EAM-guided biopsy leads to a superior diagnostic yield compared with conventional fluoroscopy-guided biopsy in patients with new-onset and persistent NICM.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. New onset NICM as defined by the presence of left ventricular dysfunction (LVEF < 45% by echocardiography and/or MRI), with symptoms or signs of HF (dyspnea, orthopnea, edema, ascites, rales or pulmonary vascular congestion on chest radiography) of less than 3 months in duration.
3. Persistent recent onset NICM as defined by the LVEF and signs/symptoms in #2 above with persistence of the LVEF < 45% despite evidence-based treatment for HF with reduced LVEF for 2 to 6 months.
4. Willingness to provide informed consent

   -

Exclusion Criteria:

1. Prior diagnosis of HF or documented LVEF < 45% more than 6 months prior to enrollment.
2. Coronary artery disease, either by history or as determined by coronary angiography demonstrating hemodynamically significant lesions deemed sufficient to potentially contribute to left ventricular dysfunction.
3. Ongoing hemodynamically significant arrhythmias deemed to be an independent cause of HF decompensation
4. Constrictive pericarditis or tamponade
5. Complex congenital heart disease
6. History of malignancy with treatment by anthracyclines or other known cardiotoxic chemotherapeutic agents
7. More than mild aortic or mitral stenosis
8. Intrinsic (prolapse, rheumatic) valve disease with severe mitral, aortic or tricuspid regurgitation
9. Primary hypertrophic cardiomyopathy
10. Untreated thyroid disease
11. Severe nutritional deficiency
12. Severe uncontrolled hypertension
13. Sepsis, active infection (excluding cystitis) or other comorbidity driving the HF decompensation
14. History of cardiac transplantation
15. Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.5 in the absence of anticoagulation treatment
16. Inability to comply with planned study procedures

    -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with New onset NICM that are scheduled for a biopsy as part of their clinical care
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy guided EMB and EAM guided EMB on all patients meeting existing guidelines for biopsy. | November 2018
  Additional biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Francis Marchlinski, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Mayo clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided